CLINICAL TRIAL: NCT01605578
Title: Description Des Populations Cellulaires Des Tissus Adipeux Sous-cutanés Abdominaux et glutéo-fémoraux Chez la Femme.
Brief Title: Description of Abdominal and Gluteo-femoral Subcutaneous Adipose Tissue Cell Population in Women - GLUTAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Basic Science
Other Study IDs: C11-48; 2011-A01496-35 (Registry Identifier: IDRCB)
Record Dates: First submitted 2012-05-11; First posted 2012-05-25 (Estimated); Last update posted 2025-09-04 (Actual); Status verified 2025-03

CONDITIONS: Adipose Tissue
MeSH Terms: interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Non-menoposal healthy volunteer women aged between 25 to 45 years (Other): Adipose tissue biopsie (2-3g) have been taken by needle biopsy form the abdomen (periumbilical) and gluteo-femoral (upper thigh) levels
  Interventions: Procedure: Biopsies

INTERVENTIONS:
Procedure: Biopsies — Abdominal and gluteo-femoral subcutaneous adipose tissue biopsies

SUMMARY:
The purpose of this study is to compare, in healthy women, the adipose tissue composition between abdomen and thigh and then determine whether differences exist independently of the state of obesity.

The findings of this study may help to explain the mechanism contributing to a beneficial role of gluteo-femoral fat contrasting with a deleterious role of abdominal fat on cardiovascular and metabolic dysfunctions.

ELIGIBILITY:
Inclusion Criteria:

* women between 15 and 45 years old
* with genital activity
* stable weight during the previous 3 months
* BMI from 20 to 28
* regular menstrual cycles (28 +/- 2 days) during the previous 3 months
* reliable means of contraception (systemic hormonal contraception, intrauterine contraceptive device, tubal ligation)
* using the same way of contraception during the previous 3 months
* normal clinical examination
* able to be compliant with the schedule of protocol assessments
* willing and able to provide written informed consent
* affiliated to a National Health Service
* agreeing to being registered on the national file for subjects participating in biomedical research

Exclusion Criteria:

* Exclusions related to significant medical disturbances :
* type I and II diabetes
* early menopause
* serious psychological disorders
* uncontrolled thyroid disorders
* know allergy to local anesthetics especially Xylocaine
* abnormal laboratory results
* medical history that, in the opinion of the investigator, makes the subject unsuitable for enrollment
* positive test result for HIV, HCV and/or HBV virus
* positive pregnancy test
* Exclusions related to subject lifestyle :
* smoking > 10 cigarettes per day
* smoking cessation during the previous 3 months
* weight fluctuation (>3kg) during the previous 3 months
* alcohol abuse
* coffee or tea consumption > 6 cups per day
* high consumption of drinks comprising xanthine bases (>0.5 liters/day)
* consumption of drinks (water or herbal teas) > 2 liters per day
* Exclusions related to previous or concomitant treatments :
* anticoagulant
* neuroleptic or antidepressant
* medication with draining, lipolytic, appetite suppressant and/or slimming effect
* local or systemic corticosteroid therapy on the test areas
* hormonal treatment other than contraception
* diuretic
* local treatment against cellulitis (mesotherapy,phosphatidylcholine injection, mechanical process)
* thighs liposuction < 2 years
* chronic treatment with anti-inflammatory
* Exclusions related to the subject :
* unwillingness or inability to comply with the requirements of the protocol
* previous participation in a clinical trial within 30 days
* inability to understand and sign the consent due to linguistic or psychic issues
* subject deprived of liberty or under guardianship, tutorship or judicial protection
* female who are currently pregnant or breastfeeding or female considering becoming pregnant while in the study

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-05-14 (Actual); Primary Completion 2012-12-14 (Actual); Study Completion 2012-12-14 (Actual)

PRIMARY OUTCOMES:
To compare the number and the phenotype of cells between abdominal and gluteo-femoral adipose tissue in women. | There is no time frame. It's a comparison of adipose tissue composition between two locations, collected both at visit 2 (inclusion).

CONTACTS AND LOCATIONS:
Overall Officials: Claire Thalamas, Doctor, Principal Investigator — CHU Purpan (Toulouse)
Locations (1):
- Centre d'Investigation Clinique, CHU Purpan, Toulouse, France

REFERENCES:
- [Background] Gao H, Volat F, Sandhow L, Galitzky J, Nguyen T, Esteve D, Astrom G, Mejhert N, Ledoux S, Thalamas C, Arner P, Guillemot JC, Qian H, Ryden M, Bouloumie A. CD36 Is a Marker of Human Adipocyte Progenitors with Pronounced Adipogenic and Triglyceride Accumulation Potential. Stem Cells. 2017 Jul;35(7):1799-1814. doi: 10.1002/stem.2635. Epub 2017 May 18. PMID 28470788